CLINICAL TRIAL: NCT03211403
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of SHR4640 in Male Subjects With High Serum Uric Acid Level
Brief Title: Multiple Doses Study of SHR4640 in Male Subjects With High Serum Uric Acid Level
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SHR4640-102-AUS
Record Dates: First submitted 2017-06-27; First posted 2017-07-07 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — ruzinurad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR4640 2.5mg (Experimental): 6 subjects assigned to 2.5mg SHR4640 and 2 subjects assigned to placebo
  Interventions: Drug: SHR4640
- SHR4640 10mg (Experimental): 6 subjects assigned to 10mg SHR4640 and 2 subjects assigned to placebo
  Interventions: Drug: SHR4640
- SHR4640 20mg (Experimental): 6 subjects assigned to 20mg SHR4640 and 2 subjects assigned to placebo
  Interventions: Drug: SHR4640

INTERVENTIONS:
Drug: SHR4640 — SHR4640 or placebo once daily for a week

SUMMARY:
This is a single-Center, randomized, double-Blind, placebo-controlled, multiple ascending-dose Phase I trail.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged between 18 and 65 years, inclusive.
2. Body weight ≥ 50 kg and body mass index between 18.0 and 35.0 kg/m2, inclusive.
3. Screening sUA level ≥0.36 mmol/L.
4. Considered generally healthy upon completion of medical history, full physical examination, vital signs, laboratory parameters (including thyroid function and serological tests, hematology, urinalysis, and biochemistry), 12-lead ECG, and abdominal ultrasound, as judged by the Investigator.
5. Agrees to use a highly effective method of contraception, i.e. condom and suitable contraception for his female partner e.g. oral contraceptive or intrauterine contraceptive device during heterosexual intercourse or be non-heterosexually active, or practice sexual abstinence throughout the study period and for 30 days following final dose of study drug, and must agree to refrain from sperm donation from Day -2 until at least 30 days following final dose of study drug.
6. Negative drug screen (including alcohol) at screening and on admission to clinical site.
7. Able to understand the study procedures and the risks involved and must be willing to provide a written informed consent before any study-related activity.

Exclusion Criteria:

1. History of hypersensitivity to SHR4640 or its analogues.
2. History of gout.
3. Screening alanine aminotransferase, aspartate aminotransferase, total bilirubin, or gamma glutamyl transferase > 1.5 × upper limit of normal.
4. Positive result for human immunodeficiency virus (HIV).
5. Positive result for hepatitis B surface antigen or hepatitis C virus antibody.
6. History or presence of kidney stones.
7. Acute or chronic illness that, in the opinion of the Investigator, might confound the results of the trial or pose risk to the subject when administering the trial product.
8. Undergone major surgery within 3 months of Day 1 or has surgery planned during study participation.
9. Donated any blood or plasma in the past month or more than 400 mL within 3 months of Day 1.
10. Has unsuitable venous for blood sampling.
11. Use of tobacco products within 30 days of Day 1.
12. Heavy caffeine drinker (more than 5 cups or glasses of caffeinated beverages per day).
13. History of drug and/or alcohol abuse in the last year.
14. Consumes more than 14 units of alcohol per week (1 unit = 250 mL beer, 25 mL of 40% spirits and 125 mL glass of wine).
15. Consumes grapefruit and/or poppy seed within 5 days of Day 1.
16. Unable to refrain from strenuous exercises, tobacco products, alcohol, grapefruit, and/or poppy seed from Day -2 to Day 10.
17. Use of any of the following, unless agreed as nonclinically relevant by the Investigator and the Sponsor:

1) Prescription medication within 2 weeks of Day 1. 2) Over-the-counter medication within 1 week of Day 1. 3) Use of any over the-counter, nutraceuticals, or prescription medications that might interfere with the absorption, distribution, metabolism, or excretion of SHR4640 (proton-pump inhibitor, fluconazole, indomethacin, ranitidine, flurbiprofen, probenecid, aprepitant, etc.) within 1 month of Day 1.

18. Received the last dose of a study drug (or treatment with a medical device) within 30 days or 5 T1/2 (whichever is longer) of the study drug of Day 1 or are currently participating in another study of a study drug (or medical device).

19. Any other medical or psychological condition, which in the opinion of the Investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements or to complete the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events in terms of changes in Hematology | Up to Day 14
  Hemoglobin Hematocrit Erythrocytes count Mean cell volume, Mean cell hemoglobin concentration, Leukocytes count, Neutrophils count, Lymphocytes count, Monocytes count, Eosinophils count, Basophils count, Platelets count
Incidence of Adverse events in terms of changes in Urinalysis | Up to Day 14
  Urobilinogen Dipstick urinalysis, including: pH, Specific gravity, Protein, Blood, Leukocytes, Glucose, Ketones, Bilirubin, Nitrites
Incidence of Adverse events in terms of changes in Biochemistry (fasting) | Up to Day 14
  Including Serum creatinine, Urea, Alanine aminotransferase, Aspartate aminotransferase, Gamma glutamyl transferase, Total bilirubin, Total protein, Albumin, Alkaline phosphatase, Serum uric acid, Glucose, Triglycerides, Total cholesterol, High-density lipoprotein cholesterol, Low-density lipoprotein cholesterol
Incidence of Adverse events in terms of changes in Physical examinations | Up to Day 14
  Review of body weight and height; general appearance; head; eyes; ears/nose/throat; neck; lymph nodes; neurological and musculoskeletal systems; heart; lungs; abdomen; skin; and extremities
Incidence of Adverse events in terms of changes in Vital signs | Up to Day 14
  Oral temperature, respiratory rate, blood pressure, and pulse rate
Incidence of Adverse events in terms of changes in 12-lead ECGs | Up to Day 14
  The 12-lead ECGs must be recorded after the subjects have rested in the supine position for 5 minutes to ensure a stable baseline.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) (of single dose and at stable status) | Up to Day 10
Area under the plasma concentration versus time curve (AUC) (of single dose and at stable status) | Up to Day 10
Half-time (T1/2) (of single dose and at stable status) | Up to Day 10
Time to the peak plasma concentration (Tmax) (of single dose and at stable status) | Up to Day 10
Changes in serum uric acid concentration from baseline | Up to Day 10
Changes in urinary uric acid excretion from baseline | Up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Sam Salman, B.Sc.BMBS, Principal Investigator — Linear Clinical Research
Locations (1):
- Atridia Pty Limited, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No